CLINICAL TRIAL: NCT00004402
Title: Phase III Randomized Study of Interferon Gamma in Children With Severe, Congenital Osteopetrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Purpose: Treatment
Other Study IDs: 199/13284; MUSC-FDR000768
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-01

CONDITIONS: Osteopetrosis
Keywords: genetic diseases and dysmorphic syndromes; osteopetrosis; rare disease
MeSH Terms: conditions — Osteopetrosis; Genetic Diseases, Inborn; Rare Diseases | interventions — Calcitriol; Interferon-gamma

INTERVENTIONS:
Drug: calcitriol
Drug: interferon gamma

SUMMARY:
OBJECTIVES: I. Compare the rate of treatment failure in osteopetrosis patients receiving interferon gamma in combination with calcitriol to the rate of treatment failure in patients receiving calcitriol alone.

II. Compare the number of adverse events or clinical manifestations of disease progression occurring in these patients.

III. Assess the effects of interferon gamma on hematopoiesis, cranial nerve function, and rate of infection in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, placebo controlled, open label study. Patients are randomized to one of two arms (interferon gamma in combination with calcitriol or calcitriol alone).

Arm I: Patients receive calcitriol once daily. Interferon gamma is administered by subcutaneous injection three times a week.

Arm II: Patients receive calcitriol once daily. Patients may continue treatment in the absence of toxicity and disease progression. If disease progression is diagnosed in the control group, patients will then receive interferon gamma in combination with calcitriol.

Patients are followed every 4 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Biopsy and x-ray confirmed primary osteopetrosis
* Presence of anemia and/or cranial nerve compression

--Prior/Concurrent Therapy--

* Biologic therapy: No prior/concurrent bone marrow transplantation No prior interferon gamma No other investigational biologic agents
* Chemotherapy: No prior/concurrent chemotherapeutic agents for bone marrow transplantation
* Endocrine therapy: Prior/concurrent corticosteroid as supportive therapy allowed
* Radiotherapy: Not specified
* Surgery: At least 5 days since major surgery
* Other: Prior/concurrent calcitriol as supportive therapy allowed Prior/concurrent transfusion as supportive therapy allowed Prior/concurrent dietary therapy allowed

--Patient Characteristics--

* Age: 2 months to 10 years
* Performance status: Not specified
* Life expectancy: At least 6 months
* Hematopoietic: Not specified
* Hepatic: Bilirubin less than 2 mg/dL
* Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 50 mL/min
* Pulmonary: No uncorrected airway obstruction
* Other: No active infection requiring intravenous antibiotics No known seizure disorder not related to hypocalcemia No uncorrected hydrocephalus No MRI evidence of cerebral atrophy Must maintain or gain body weight No sleep apnea No thrombocytopenia No massive splenomegaly

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 1999-11; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: L. Lyndon Key, Jr., Study Chair — Medical University of South Carolina